CLINICAL TRIAL: NCT00790920
Title: A Randomised, Double-blind, Parallel-group Placebo-controlled Phase III Study to Evaluate the Efficacy and Safety of Desmoteplase in Subjects With Acute Ischemic Stroke
Brief Title: Efficacy and Safety Study of Desmoteplase to Treat Acute Ischemic Stroke
Acronym: DIAS-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12402A; 2008-000622-40 (EudraCT Number)
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Stroke
Keywords: Acute ischemic stroke; Angiography; Desmoteplase; Thrombolytic
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — salivary plasminogen activator alpha 1, Desmodus rotundus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Desmoteplase (Experimental)
  Interventions: Drug: Desmoteplase
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desmoteplase — 90 μg/kg bodyweight, IV, single bolus over 1 - 2 minutes on 1st day
  Arms: Desmoteplase
Drug: Placebo — IV, single bolus over 1 - 2 minutes on 1st day
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether desmoteplase is effective and safe in the treatment of patients with acute ischaemic stroke when given within 3-9 hours from onset of stroke symptoms.

DETAILED DESCRIPTION:
Acute stroke is a major cause of mortality and long-term disability in the developed world. The only currently approved thrombolytic intervention for acute ischemic stroke, which constitutes the majority of strokes, is alteplase (recombinant tissue plasminogen activator; rtPA). The use of alteplase is limited as it is approved for use within 3 hours after symptom onset and by the risk of inducing intracerebral haemorrhage; consequently fewer than 3% of acute stroke subjects are treated. The thrombolytic agent desmoteplase (recombinant Desmodus Salivary Plasminogen Activator alpha-1; rDSPAalpha-1) produced by recombinant biotechnology has its naturally occurring counterpart in the saliva of the vampire bat Desmodus rotundus. Compared to alteplase, desmoteplase has a more favourable profile in terms of high fibrin specificity and non neurotoxicity.

The study aims to confirm efficacy and safety of desmoteplase for thrombolytic therapy of patients with acute ischaemic stroke in the extended time window of 3-9 hours after onset of stroke symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute ischemic stroke
* Informed consent
* Age between 18 and 85 years
* Treatment can be initiated within 3-9 hours after the onset of stroke symptoms
* NIHSS Score of 4-24
* Vessel occlusion or high-grade stenosis on MRI or CTA in proximal cerebral arteries

Exclusion Criteria:

* Pre-stroke mRS >1
* Previous exposure to desmoteplase
* Extensive early infarction on MRI or CT in any affected area
* Imaging evidence of ICH or SAH; AV malformation; cerebral aneurysm; or cerebral neoplasm
* Internal carotid artery occlusion on the side of the stroke lesion
* Treatment with heparin in the past 48 hours and a prolonged partial thromboplastin time
* Treatment with oral anticoagulants and a prolonged prothrombin time
* Treatment with glycoprotein IIb - IIIa inhibitors within the past 72 hours. Use of single agent oral platelet inhibitors is permitted
* Treatment with a thrombolytic agent within the past 72 hours

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2008-12; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale Score | 90 days

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) Score | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (102):
- Australia (6):
  - AU006, Clayton
  - AU004, Gosford
  - AU001, Melbourne
  - AU002, Melbourne
  - AU003, Newcastle
  - AU009, Perth
- Austria (5):
  - AT003, Graz
  - AT004, Innsbruck
  - AT002, Linz
  - AT001, Linz
  - AT005, Vienna
- Estonia (4):
  - EE002, Tallinn
  - EE004, Tallinn
  - EE003, Tallinn
  - EE001, Tartu
- France (12):
  - FR004, Besançon
  - FR013, Bordeaux
  - FR003, Bourg-en-Bresse
  - FR015, Caen
  - FR014, Lille
  - FR012, Limoges
  - FR008, Montpellier
  - FR010, Nice
  - FR001, Paris
  - FR009, Paris
  - FR007, Perpignan
  - FR016, Toulouse
- Germany (13):
  - DE002, Berlin
  - DE001, Dresden
  - DE011, Erlangen
  - DE005, Freiburg im Breisgau
  - DE018, Hamburg
  - DE020, Hanover
  - DE019, Jena
  - DE003, Leipzig
  - DE022, Lübeck
  - DE021, Neuruppin
  - DE025, Rostock
  - DE012, Schweinfurt
  - DE016, Würzburg
- Hong Kong (2):
  - HK001, Hong Kong
  - HK002, Hong Kong
- India (6):
  - IN004, Chandigarh
  - IN009, Guntur
  - IN008, Hyderabad
  - IN003, Hyderabad
  - IN007, Ludhiana
  - IN001, Pune
- Netherlands (2):
  - NL001, Breda
  - NL002, Groningen
- Philippines (3):
  - PH003, Manila
  - PH001, Pasig
  - PH002, Quezon City
- Poland (5):
  - PL004, Gdansk
  - PL005, Lublin
  - PL006, Sandomierz
  - PL001, Warsaw
  - PL002, Warsaw
- Singapore (2):
  - SG002, Singapore
  - SG001, Singapore
- South Korea (13):
  - KR013, Ansan-si
  - KR003, Anyang
  - KR006, Busan
  - KR011, Daegu
  - KR002, Incheon
  - KR010, Kwangju
  - KR008, Seongnam
  - KR004, Seoul
  - KR001, Seoul
  - KR012, Seoul
  - KR009, Seoul
  - KR005, Seoul
  - KR007, Wŏnju
- Spain (11):
  - ES010, Albacete
  - ES012, Alcázar de San Juan
  - ES007, Barcelona
  - ES003, Barcelona
  - ES014, Bilbao
  - ES004, Girona
  - ES013, Lugo
  - ES011, Madrid
  - ES005, Madrid
  - ES008, Madrid
  - ES006, Valladolid
- CH001, Lausanne, Switzerland
- Taiwan (9):
  - TW003, Kaohsiung City
  - TW001, Kaohsiung City
  - TW006, Taichung
  - TW005, Tainan
  - TW008, Tainan
  - TW009, Taipei
  - TW007, Taipei
  - TW002, Taipei
  - TW004, Taoyuan District
- Thailand (6):
  - TH003, Bangkok
  - TH002, Bangkok
  - TH006, Bangkok
  - TH004, Bangkok
  - TH005, Chiang Mai
  - TH001, Pathum Thani
- Vietnam (2):
  - VN002, Hanoi
  - VN001, Ho Chi Minh City

REFERENCES:
- [Derived] Albers GW, von Kummer R, Truelsen T, Jensen JK, Ravn GM, Gronning BA, Chabriat H, Chang KC, Davalos AE, Ford GA, Grotta J, Kaste M, Schwamm LH, Shuaib A; DIAS-3 Investigators. Safety and efficacy of desmoteplase given 3-9 h after ischaemic stroke in patients with occlusion or high-grade stenosis in major cerebral arteries (DIAS-3): a double-blind, randomised, placebo-controlled phase 3 trial. Lancet Neurol. 2015 Jun;14(6):575-84. doi: 10.1016/S1474-4422(15)00047-2. Epub 2015 Apr 30. PMID 25937443
- See also: EMA EudraCT Result Posting — https://www.clinicaltrialsregister.eu/ctr-search/trial/2008-000622-40/results